CLINICAL TRIAL: NCT00731367
Title: A Phase IIIb, Randomized Comparative Evaluation of Two AQUACEL Ag Protocols of Care for the Management of Donor Sites.
Brief Title: Comparative Evaluation of Two AQUACEL Ag Protocols of Care for the Management of Donor Sites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Daniel Caruso, Arizona Burn Center, Maricopa Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CW-0412-05-A080
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Split-Thickness Donor Sites.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gelled (Active Comparator): Aquacel Ag gelled.
  Interventions: Device: Aquacel Ag Gelled
- Adherent (Active Comparator): Aquacel Ag adherent
  Interventions: Device: Aquacel Ag Adherent

INTERVENTIONS:
Device: Aquacel Ag Gelled — AQUACEL Ag is produced by changing a small fraction of the sodium ions present in AQUACEL for silver ions and then stabilizing the complex formed by adding chloride. This produces a characteristic silver gray product. There are no counter ions (such as nitrate or sulphadiazine ions) present: these compounds, found in many silver containing products, are known to retard wound healing. AQUACEL Ag maintains a moist wound-healing environment while, at the same time, killing wound pathogens that are immobilized within the dressing. It also reduces bioburden at the wound-dressing surface, thus minimizing the risk of wound infection and facilitating wound healing.
  Arms: Gelled
Device: Aquacel Ag Adherent — AQUACEL Ag is produced by changing a small fraction of the sodium ions present in AQUACEL for silver ions and then stabilizing the complex formed by adding chloride. This produces a characteristic silver gray product. There are no counter ions (such as nitrate or sulphadiazine ions) present: these compounds, found in many silver containing products, are known to retard wound healing. AQUACEL Ag maintains a moist wound-healing environment while, at the same time, killing wound pathogens that are immobilized within the dressing. It also reduces bioburden at the wound-dressing surface, thus minimizing the risk of wound infection and facilitating wound healing.
  Arms: Adherent

SUMMARY:
This phase IIIb, randomized, comparative, multi-center study is designed to evaluate two AQUACEL Ag protocols of care for the management of split-thickness donor sites. Both protocols of care will utilize AQUACEL Ag as the primary dressing. As per the randomization assignment, one protocol of care will have the AQUACEL Ag initially covered with a gauze dressing to create an adherent state and in the other protocol of care the AQUACEL Ag will be covered with a transparent film to maintain a gelled state.

The primary objective of the study will be to quantify the proportion of subjects healed at 14 days. Secondary objectives will include: time to healing, degree of pain at dressing change and while wearing the dressing, simplicity of use, resources used in treatment and safety. Approximately 68 subjects will be enrolled from 10 centers from within the US and Canada.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative must provide written informed consent.
* Subject who is younger than legal consenting age must have a legally authorized representative who will provide written informed consent.
* The subject is scheduled to undergo a split-thickness skin graft (autograft)
* Harvesting of the donor site must be limited to the location and size of the anterior thigh
* The selected anterior thigh must be a first - time harvesting.

Exclusion Criteria:

* Subjects with known skin sensitivity to any of the dressing components.
* Subjects who require a full thickness graft.
* The subject with a poor prognosis, which would make it unlikely that he/she would survive the 21 day study period.
* Subjects who have been previously randomized into the study, or who are presently participating in another clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the proportion of subjects healed. | 14 days

SECONDARY OUTCOMES:
Time to healing. | 14 days
Degree of pain at dressing change. | 14 days
Degree of pain/discomfort while wearing the dressing at rest and during mobility. | 14 days
Investigator's rating of dressing performance (per subject and overall). | 14 days
Resources utilization. | 14 days
Readiness for re-harvesting. | day 14
Safety. | 14 days +30

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Caruso, MD, Principal Investigator — Maricopa Medical Center
Locations (1):
- Maricopa Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Sinha S, Gabriel VA, Arora RK, Shin W, Scott J, Bharadia SK, Verly M, Rahmani WM, Nickerson DA, Fraulin FO, Chatterjee P, Ahuja RB, Biernaskie JA. Interventions for postburn pruritus. Cochrane Database Syst Rev. 2024 Jun 5;6(6):CD013468. doi: 10.1002/14651858.CD013468.pub2. PMID 38837237
- [Derived] Blome-Eberwein S, Johnson RM, Miller SF, Caruso DM, Jordan MH, Milner S, Tredget EE, Sittig KM, Smith L. Hydrofiber dressing with silver for the management of split-thickness donor sites: a randomized evaluation of two protocols of care. Burns. 2010 Aug;36(5):665-72. doi: 10.1016/j.burns.2009.06.193. Epub 2009 Dec 6. PMID 19969423